CLINICAL TRIAL: NCT03745443
Title: The Assessment of Efficacy and Safety of Step-wise up and Down PEEP Titration in Healthy Pediatric Patients Under General Anesthesia
Brief Title: Efficacy of Recruitment Maneuver in Pediatric Patients Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mother and Child Health Institute of Serbia Dr Vukan Cupic (Other)
Responsible Party: Principal Investigator, Ana Mandras, Principal Investigator Anesthesiologist, Mother and Child Health Institute of Serbia Dr Vukan Cupic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8/30,2017
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Healthy
MeSH Terms: interventions — Ventilation

STUDY DESIGN:
Intervention Model Description: randomized parallel controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention: increase and decrease positive end-expiratory pressure. PEEP titration: 20 minutes before the end of anesthesia and surgery PEEP was increased by 2 on every 5 breaths to 11 ventilation was maintained on PEEP 11 for 2 minutes.Then, PEEP was reduced by 2 for every 5 breaths to 5.Total time to titrate was 5 minutes.
  Interventions: Procedure: increase and decrease positive end-expiratory pressure
- Control (No Intervention): Ventilation with PEEP 3 during anesthesia and surgery

INTERVENTIONS:
Procedure: increase and decrease positive end-expiratory pressure — 20 minutes before the end of anesthesia and surgery PEEP was increased by 2 on every 5 breaths to 11. Ventilation with PEEP 11 was maintained for 2 minutes. Then, PEEP was reduced by 2 on every 5 breaths to 5 cmH2O
  Other Names: ventilation with PEEP 3
  Arms: Intervention group

SUMMARY:
During general anesthesia lung collapses and atelectasis occurs. Preservation of atelectasis can cause pulmonary disfunction. The goal of safe anesthesia is to protect the lungs intraoperatively. Positive end-expiratory pressure (PEEP) is distending pressure that prevents alveolar collapse during mechanical ventilation and is a part of recruitment maneuver that is often used in patients on mechanical ventilation. Overall effect of PEEP is improvement in lung function. PEEP can have adverse effects on hemodynamics. The objective of this study was to assess the effect of step up and down PEEP titration on lung function and hemodynamics in healthy preschool children during general anesthesia. One group of children was ventilated with constant PEEP. the other was submitted to PEEP titration. Changes in lung compliance, gas exchange and hemodynamic status were documented as well as any unwanted effects.

DETAILED DESCRIPTION:
Seventy preschool children American Society of Anesthesiologists classification system (ASA) I and II scheduled for non-cardiothoracic surgery were allocated in two groups. Interventional group (n=35) received PEEP titration and Control group (n=35) didn't. They were ventilated only with PEEP 3. PEEP titration: In Intervention group, 20 minutes before the end of anesthesia PEEP was increased by 2 on every 5 breaths to 11. Ventilation with PEEP 11 was maintained for 2 minutes. Then PEEP was reduced by 2 on every 5 breaths to 5 and remain as until awakening. Total time to perform titration was 5 minutes. Blood was collected in both groups, in equal points of time that is: after induction, 20 minutes before the end of surgery and after the end of surgery (20th minute). Investigators tested differences of outcome variables between groups and within the Interventional group before and after PEEP titration. Hemodynamic monitoring and monitoring of lung function were conducted in Interventional group to observe changes during PEEP titration.

ELIGIBILITY:
Inclusion Criteria:

* age 3-7; ASA I and II
* absence of cardiovascular and respiratory comorbidity

Exclusion criteria:

* current or recent (up to 4 weeks) upper airway infection
* present of gastroesophageal reflux
* allergic reactions to anesthetics
* contraindication to chosen anesthetics

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Partial pressure of oxygen | 10 minutes after PEEP titration
  measured partial pressure of oxygen in arterial blood at the end of surgery in Interventional and Control group.
Partial pressure of carbon dioxide | 10 minutes after PEEP titration
  measured partial pressure carbon dioxide in arterial blood at the end of surgery in Interventional and in Control group
Lung compliance | 10 minutes after PEEP titration
  spirometric measurement of dynamic lung compliance at the end of surgery in Interventional and Control group
Lung compliance | 5 minutes
  spirometric measurement of dynamic lung compliance on different PEEP levels in Interventional group

SECONDARY OUTCOMES:
postoperative hemoglobin oxygen saturation | 4 hours after extubation
  hemoglobin oxygen saturation measured with puls oximeter
intraoperative hemodynamic status | 5 minutes
  invasive blood pressure monitoring during PEEP titration in Interventional group
intraoperative respiratory adverse effect | 5 minutes
  airway pressure monitoring during PEEP titration in Interventional group

CONTACTS AND LOCATIONS:
Overall Officials: Ana Mandras, MD, Principal Investigator — Institute for Mother and Child Health Care
Locations (1):
- Institute for Mother and Child Health Care dr Vukan Cupic, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doras C, Le Guen M, Petak F, Habre W. Cardiorespiratory effects of recruitment maneuvers and positive end expiratory pressure in an experimental context of acute lung injury and pulmonary hypertension. BMC Pulm Med. 2015 Jul 31;15:82. doi: 10.1186/s12890-015-0079-y. PMID 26228052
- [Background] Boriosi JP, Sapru A, Hanson JH, Asselin J, Gildengorin G, Newman V, Sabato K, Flori HR. Efficacy and safety of lung recruitment in pediatric patients with acute lung injury. Pediatr Crit Care Med. 2011 Jul;12(4):431-6. doi: 10.1097/PCC.0b013e3181fe329d. PMID 21057351
- [Background] Cruces P, Gonzalez-Dambrauskas S, Cristiani F, Martinez J, Henderson R, Erranz B, Diaz F. Positive end-expiratory pressure improves elastic working pressure in anesthetized children. BMC Anesthesiol. 2018 Oct 24;18(1):151. doi: 10.1186/s12871-018-0611-8. PMID 30355345
- [Result] Mascotto G, Bizzarri M, Messina M, Cerchierini E, Torri G, Carozzo A, Casati A. Prospective, randomized, controlled evaluation of the preventive effects of positive end-expiratory pressure on patient oxygenation during one-lung ventilation. Eur J Anaesthesiol. 2003 Sep;20(9):704-10. doi: 10.1017/s0265021503001145. PMID 12974591